CLINICAL TRIAL: NCT06385405
Title: Repetitive Transcranial Magnetic Stimulation(rTMS) Treatment Based on Personalized Modulation of Electroencephalography Promotes Symptom Remission in Major Depressive Disorder (MDD) - A Randomized Controlled Clinical Trial
Brief Title: Electroencephalography-based Precise Repetitive Transcranial Magnetic Stimulation Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Shanghai Municipal Science and Technology Commission (Other Government); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, Professor, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024y0423
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Transcranial magnetic stimulation(TMS); electroencephalogram (EEG); Personalized treatment; machine learning
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: To test the hypothesis that repetitive transcranial magnetic stimulation based on individualized EEG modulation may be more effective in promoting symptomatic relief of major depressive disorder (MDD), patients were tested in a parallel controlled trial.During the treatment period, patients will be randomly grouped into the precision group, which will be treated with rTMS based on personalized modulation of EEG data, and the conventional group, which will be treated with TMS at a frequency of 10 Hz to stimulate the left dorsolateral prefrontal cortex (DLPFC).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Precision Group (Experimental): Patients in the precision group will be treated with Individualized alpha frequency Transcranial Magnetic Stimulation (αTMS) Treatment.
  Interventions: Device: Individualized alpha frequency Transcranial Magnetic Stimulation (αTMS) Treatment
- The Conventional Group (Active Comparator): Patients in the conventional group will be treated with 10Hz-frequency TMS over the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: 10Hz-frequency TMS treatment over the left dorsolateral prefrontal cortex (DLPFC)

INTERVENTIONS:
Device: Individualized alpha frequency Transcranial Magnetic Stimulation (αTMS) Treatment — The target site for alpha frequency Transcranial Magnetic Stimulation (αTMS) was identified based on alterations in alpha band spectral connectivity, which were measured using four frontal electroencephalography (EEG) channels (F1, F3, F5, FC3) subsequent to 10Hz transcranial magnetic stimulation (TMS). Alpha band spectral connectivity refers to the degree of similarity between the spectral waveforms of the alpha band across channels. The alpha frequency stimulation rate was defined as the highest spectral peak within the alpha band ranging from 7 to 13 Hz of the target channel. Each treatment cycle consisted of 20 daily sessions over a 4-week span, and stimulation was administered for 2 seconds every minute for a total duration of 20 minutes at 80% of the individual's motor threshold.
  Arms: The Precision Group
Device: 10Hz-frequency TMS treatment over the left dorsolateral prefrontal cortex (DLPFC) — Prefrontal Transcranial Magnetic Stimulation (TMS) therapy repeated daily over 4 weeks (20 sessions) is US Food and Drug Administration (FDA) approved for treating Major Depressive Disorder in adults who have not responded to prior antidepressant medications. The strongest evidence supports high-frequency treatment over the left dorsolateral prefrontal cortex (DLPFC). The common stimulation frequency is 10Hz. It is usually applied for a duration of 4 weeks, 5 days a week.
  Arms: The Conventional Group

SUMMARY:
This study will focus on the hypothesis that repetitive transcranial magnetic stimulation (TMS) based on EEG personalized modulation may be more effective in promoting symptomatic relief of major depressive disorder (MDD), and will rely on the platform of neuroimaging and function brain imaging of Shanghai Mental Health Center (SMHC), an authoritative institution in the field of mental health. We will eventually facilitate optimization of physical therapy for major depressive disorder (MDD).

DETAILED DESCRIPTION:
Major depression disorder (MDD) is increasingly conceptualized as a disorder of brain networks, which related to dysregulation of functional connectivity. rTMS has the advantages of being safe, non-invasive and well-tolerated, and has been clarified by the FDA to be used in the treatment of depression with some positive efficacy. Machine learning based on EEG data, exploring machine learning and big data analytics methods, and applying the output reference value recommendations to the personalized treatment of depressed patients are expected to be more effective in promoting the alleviation of patients' depressive symptoms.

Every participant meeting the inclusion criteria will be fully informed of the study and be asked to sign the written informed consent before enrollment. Outpatient physicians will conduct the initial screening, collecting all diagnostic and medication information from the medical records at each follow-up visit. Several psychiatrists, all of whom are qualified and well-trained, will conduct clinical assessments at baseline and follow-up at the end of weekly TMS treatments, as well as clinical follow-up 3 months after the end of treatment. Clinical assessments will include HAMD, HAMA, CGI scale and etc. EEG parameter assessments will include changes in alpha-band spectral connectivity at baseline and after every 5 TMS treatments.

During the treatment period, patients will be randomly grouped into the precision group, which will be treated with rTMS based on personalized modulation of EEG data, and the conventional group, which will be treated with TMS at a frequency of 10 Hz to stimulate the left dorsolateral prefrontal cortex (DLPFC). The treatments will be administered once a day, 5 times a week for 4 weeks, totaling 20 sessions. At the end of each week's treatment the patient's EEG will be recorded and the patient will be clinically evaluated by a qualified and well-trained psychiatrist. The original medication regimen will be maintained as much as possible during the treatment period, and adverse effects such as headaches will be faithfully recorded.

The sample size calculation for this study was based on a priori power analysis using G*Power 3.1.9.7. Among the imputed parameters it was chosen to include α = 0.05, power (1-ß) = 0.9. We used effect size f = 0.2 as parameter for the effect size estimation, based on the findings from previous study reported that the depressive symptom changes before and after rTMS intervention in patients with MDD. Two groups, corresponding to the two experimental conditions of the study, and age, sex, educational level, symptom, in total of 4 covariates were included. Taking into account a dropout rate of 15%, the final estimated number of participants is 70.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of participants should be made in accordance to the diagnostic criteria described for Major Depressive Disorder (MDD) of the Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-V).
* be willing to receive neuromodulation therapy and sign the written informed consent
* an age of 16-65 years
* The patient's medication regimen is based on only one antidepressant, and the medication regimen is not adjusted as much as possible during the treatment period.
* Having a total score of not less than 20 on the Hamilton Depression Rating Scale (HAMD-24).
* sufficient hearing or reading ability

Exclusion Criteria:

* History of electroconvulsive therapy (ECT)
* Presence of metallic foreign bodies near the stimulation coil or stimulation scalp, e.g., intracranial metal implants, cochlear implants, built-in pulse generators (brain pacemakers, cardiac pacemakers)
* Epilepsy
* Pregnancy
* History of head injury
* Mental disorders such as schizophrenia, bipolar disorder, schizoid personality disorder, alcohol/drug abuse or dependence, etc.
* Serious physical illnesses
* Taking medication that lowers the seizure threshold
* Participating in any clinical trial within 30 days before the baseline
* Other situations judged by the investigators not to be suitable for the clinical trial

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
the response rate | 4 weeks
  It will be determined by Hamilton Depression Scale(HAMD-24 item) score. Specifically, the response rate is defined as a 30% decrease in HAMD score from those measured at baseline.

SECONDARY OUTCOMES:
complete remission rate | 4 weeks
  It will be determined by Hamilton Depression Scale(HAMD-24 item) score. Specifically, the complete remission rate is defined as the HAMD score of less than 8 at the follow-up point.
alpha band spectral connectivity in electroencephalogram (EEG) parameters | 4 weeks
  It will be determined by the changes of alpha band spectral connectivity in EEG parameters. Specifically, the EEG index is the change in alpha band spectral connectivity before and after a single TMS intervention, representing the functional connectivity between the frontal lobe and other brain regions across the entire brain.
Evaluation of therapeutic effect | 4 weeks
  It will be determined using the criteria for the global improvement(GI) from Clinical Global Impression(CGI). Specifically, the global improvement(GI) will be rated by the clinician for the degree of improvement in the subject's current condition compared to baseline at enrollment on an 8-point scale from 0-7(the rating "1" refers to significant progress, and the rating "2" refers to progress, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: TianHong Zhang, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No